CLINICAL TRIAL: NCT05777369
Title: An Open, Single-arm, Multicenter Study of R-CMOP Protocol for Primary Treatment of Diffuse Large B-cell Lymphoma Based on Cardiac Function Screening
Brief Title: R-CMOP in Patients With Primary Diffuse Large B-cell Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DED-DLBCL-K08
Record Dates: First submitted 2023-03-09; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: DLBCL; R-CMOP; Mitoxantrone liposome
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Cyclophosphamide; Vincristine; Vindesine; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- R-CMOP (Experimental): R-CMOP：Rituximab, Cyclophosphamide, Mitoxantrone hydrochloride liposomes, Vincristine or Vindesine, Prednisone
  Interventions: Drug: Rituximab; Drug: Mitoxantrone hydrochloride liposome; Drug: Cyclophosphamide; Drug: Vincristine/Vindesine; Drug: Prednisone

INTERVENTIONS:
Drug: Rituximab — 375 mg/m2, d0
Drug: Mitoxantrone hydrochloride liposome — 18 mg/m2, d1
Drug: Cyclophosphamide — 750 mg/m2, d1
Drug: Vincristine/Vindesine — Vincristine: 1.4 mg/m2, d1(The maximum dose was 2 mg) Vindesine: 3 mg/m2, d1
Drug: Prednisone — 60 mg/m2, d1~d5

SUMMARY:
To evaluate the efficacy and safety of R-CMOP regimen based on mitoxantrone hydrochloride liposome injection in the treatment of newly diagnosed diffuse large B-cell lymphoma (DLBCL) based on cardiac function screening

DETAILED DESCRIPTION:
Compared with traditional mitoxantrone, mitoxantrone liposomes can significantly prolong the survival time of patients and reduce the cardiotoxicity and non-hematological toxicity of anthracycline drugs. Based on the cardiac safety and efficacy of mitoxantrone liposome, the R-CMOP scheme based on Mitoxantrone liposome for the treatment of initial DLBCL based on cardiac function screening has sufficient theoretical basis and is worth exploring.

ELIGIBILITY:
Inclusion Criteria:

1. To participate in the study voluntarily and sign the informed consent (ICF);
2. 18 years ≤ age ≤80 years;
3. Expected survival time ≥3 months;
4. Initial DLBCL confirmed by histopathology;
5. There must be at least one evaluable or measurable lesion in line with Lugano2014 criteria: lymph node lesion, the length and diameter of detectable lymph node must be greater than 1.5cm; For non-lymph node lesions, the diameter of extrinsic lesions should be > 1.0cm;
6. ECOG score 0~2;
7. Bone marrow function: neutrophil count ≥1.5×10^9/L, platelet count ≥75×10^9/L, hemoglobin ≥80 g/L (neutrophil count ≥1.0×10^9/L, platelet count ≥50×10^9/L, hemoglobin ≥75g/L in patients with bone marrow involvement);
8. Liver and kidney function: serum creatinine ≤1.5 times the upper limit of normal value; AST and ALT ≤2.5 times the upper limit of normal value (≤5 times the upper limit of normal value for patients with liver invasion); Total bilirubin ≤1.5 times the upper limit of normal value (≤3 times the upper limit of normal value for patients with liver invasion);
9. Cardiac function: 50% ≤ LVEF ≤ 55%, or LVEF>55% patients with cardiovascular disease (including left ventricular enlargement (left ventricular diameter: male>60mm; female>55mm), controllable arrhythmia (first degree atrioventricular block, second degree type I atrioventricular block, atrial fibrillation, atrial flutter, ventricular premature beats (<4000 times/24h, mainly single)), myocarditis, pericarditis, structural heart disease, etc.).

Exclusion Criteria:

1. Hypersensitivity to any study drug or its components;
2. Uncontrollable systemic diseases (such as progressive infection, uncontrollable hypertension, diabetes, etc.);
3. Cardiac function and disease conform to one of the following conditions:

   1. Long QTc syndrome or QTc interval >480 ms;
   2. Complete left bundle branch block, complete right bundle branch block with left anterior branch block, second degree type II, or third degree atrioventricular block;
   3. New York College of Cardiology Grade ≥ III;
   4. A history of acute myocardial infarction, unstable angina pectoris, severely unstable ventricular arrhythmias or any other arrhythmia requiring treatment, a history of clinically severe pericardial disease, or electrocardiographic evidence of acute ischemic or active conduction abnormalities within the 6 months prior to treatment.
4. Hepatitis B and hepatitis C active infection (hepatitis B virus surface antigen positive and hepatitis B virus DNA more than 1x10^4 copies /mL; HCV RNA over 1x10^4 copies /mL);
5. Human immunodeficiency virus (HIV) infection (HIV antibody positive);
6. Past or present co-existing malignancies (other than non-melanoma basal cell carcinoma of the skin, carcinoma in situ of the breast/cervix, and other malignancies that have been effectively controlled without treatment in the past five years);
7. Had primary or secondary central nervous system (CNS) lymphoma or had a history of CNS lymphoma at the time of recruitment
8. Pregnant and lactating women and patients of childbearing age who do not want to take contraceptive measures;
9. Other researchers judged that it was not suitable to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | up to 6 cycles of chemotherapy (each cycle is 21 days)
  Objective response rate (ORR) after 6 cycles of R-CMOP chemotherapy

SECONDARY OUTCOMES:
Complete remission rate(CRR) | up to 6 cycles of chemotherapy (each cycle is 21 days)
  Complete remission rate(CRR) after 6 cycles of R-CMOP chemotherapy
Duration of remission(DOR) | up to 6 cycles of chemotherapy (each cycle is 21 days)
  Time from reaching CR or PR for the first time to disease progression
Progression-Free-Survival rate | 1 year
  from date of inclusion to date of progression, relapse, or death from any cause
Overall survival rate | 1 year
  from the date of inclusion to date of death, irrespective of cause
Adverse events (AE) | From the first day of medication to 28 days after the last dose
  The safety of the drug was evaluated by NCI-CTC AE 5.0 standard

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xu, PhD& MD, Principal Investigator — The first Affiliated Hospital Of Nanjing Medical University(JiangSu Province Hospital)